CLINICAL TRIAL: NCT02704572
Title: Comparison of Immune Response Induced by Zoster Vaccine According to the Timing of Vaccination After Zoster Illness
Brief Title: Optimal Timing of Zoster Vaccine After Zoster Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Wan Beom Park, Associate Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H1511046718
Record Dates: First submitted 2016-03-01; First posted 2016-03-10 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Shingles
Keywords: Herpes zoster vaccine; cell-mediated immunity
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6months to 2years after shingles (Experimental): Patients will be vaccinated with Zostavax from 6 months to 2 years after zoster illness.
  Interventions: Biological: Zostavax
- 2years to 5years after shingles (Active Comparator): Patients will be vaccinated with Zostavax from 2 years to 5 years after zoster illness.
  Interventions: Biological: Zostavax

INTERVENTIONS:
Biological: Zostavax — Zostavax will be administrated by subcutaneous injection.

SUMMARY:
The purpose of this study is to determine the optimal timing of zoster vaccination to induce both higher cell-mediated immunity and humoral immunity in adult patients aged over 50 with history of zoster within 5 years.

DETAILED DESCRIPTION:
Zoster vaccination is recommended by FDA for adults aged 60 years or older, and is approved for people aged 50 through 59 years old. For patients who had shingles, there is no specific length of time they must wait before receiving shingles vaccine. It is generally recommended that patients should wait for 6 to 12 months after recovery.

The investigators plan to make scientific recommendation for optimal timing of zoster vaccine after zoster illness by comparing immune response between two groups (vaccination at 6 months to 2 years after shingles vs. 2 to 5 years after shingles). Primary outcome is ELISPOT response at week 6 after vaccination. Secondary outcome is gpELISA titer at week 6 after vaccination.

All the patients will be asked if they have any contraindications for zoster vaccine by a physician before vaccination. And they will be monitored for any adverse reaction of the vaccination after 6 weeks (visiting the hospital).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50 years or older who have had shingles in 5 years
* Adults who did not receive zoster vaccination yet
* Adults who can understand and agreed with the informed consents.

Exclusion Criteria:

* Adults who have conditions which is contraindication for zoster vaccine
* Adults who had zoster vaccination already
* Adults who take immunosuppressants
* Human Immunodeficiency Virus (HIV) patients whose CD4 T cell counts below 500/mm3
* Adults with autoimmune disease who are anticipated to have a problem with immunogenicity for vaccine
* Adults who had organ transplantation and receive immunosuppressants
* Adults who are suspected to have active infectious disease
* Adults who are not eligible for zoster vaccination by investigator's assessment

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Varicella-zoster virus-specific interferon-gamma ELISPOT response | before Zostavax vaccination and at week 6 after vaccination
  Investigators measure the number of SFC (spot forming cells) using interferon-gamma ELISPOT (enzyme-linked immunospot) assay at both right before vaccination and week 6 after vaccination and see the change between two values.

SECONDARY OUTCOMES:
Antibody titer against glycoprotein of varicella-zoster virus | before Zostavax vaccination and at week 6 after vaccination
  Investigators measure the titer of VZV-specific glycoprotein-based enzyme-linked immunosorbent assay at both right before vaccination and week 6 after vaccination and see the fold change between two values.

CONTACTS AND LOCATIONS:
Overall Officials: Wan Beom Park, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gilbert PB, Gabriel EE, Hudgens MG, Miao X, Li X, Su SC, Parrino J, Chan IS. Reply to Dunning. J Infect Dis. 2015 Nov 1;212(9):1521-3. doi: 10.1093/infdis/jiv287. Epub 2015 May 17. No abstract available. PMID 25985906
- [Background] Levin MJ, Oxman MN, Zhang JH, Johnson GR, Stanley H, Hayward AR, Caulfield MJ, Irwin MR, Smith JG, Clair J, Chan IS, Williams H, Harbecke R, Marchese R, Straus SE, Gershon A, Weinberg A; Veterans Affairs Cooperative Studies Program Shingles Prevention Study Investigators. Varicella-zoster virus-specific immune responses in elderly recipients of a herpes zoster vaccine. J Infect Dis. 2008 Mar 15;197(6):825-35. doi: 10.1086/528696. PMID 18419349
- [Background] Mills R, Tyring SK, Levin MJ, Parrino J, Li X, Coll KE, Stek JE, Schlienger K, Chan IS, Silber JL. Safety, tolerability, and immunogenicity of zoster vaccine in subjects with a history of herpes zoster. Vaccine. 2010 Jun 7;28(25):4204-9. doi: 10.1016/j.vaccine.2010.04.003. Epub 2010 Apr 21. PMID 20416263
- [Background] Kim JW, Min CK, Mun YC, Park Y, Kim BS, Nam SH, Koh Y, Kwon JH, Choe PG, Park WB, Kim I. Varicella-zoster virus-specific cell-mediated immunity and herpes zoster development in multiple myeloma patients receiving bortezomib- or thalidomide-based chemotherapy. J Clin Virol. 2015 Dec;73:64-69. doi: 10.1016/j.jcv.2015.10.018. Epub 2015 Oct 24. PMID 26546878
- [Background] Kang CI, Choi CM, Park TS, Lee DJ, Oh MD, Choe KW. Incidence of herpes zoster and seroprevalence of varicella-zoster virus in young adults of South Korea. Int J Infect Dis. 2008 May;12(3):245-7. doi: 10.1016/j.ijid.2007.08.002. Epub 2007 Oct 18. PMID 17950022
- [Derived] Lee E, Chun JY, Song KH, Choe PG, Bang JH, Kim ES, Kim HB, Park SW, Kim NJ, Park WB, Oh MD. Optimal Timing of Zoster Vaccination After Shingles: A Prospective Study of the Immunogenicity and Safety of Live Zoster Vaccine. Infect Chemother. 2018 Dec;50(4):311-318. doi: 10.3947/ic.2018.50.4.311. PMID 30600654